CLINICAL TRIAL: NCT00704977
Title: Evaluation of Alcohol 20% for Separation of Pterygium Tissue During Pterygium Surgery and Comparison of Three Different Methods of Wound Closure in Pterygium Surgery: Bare Sclera, Sliding Flap, Amniotic Membrane With Biological Glue
Brief Title: Alcohol 20% for Separation of Pterygium and Comparison of Different Wound Closure Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Prof Tova Lifshitz, Soroka university Medical center, chief of ophthalmology department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor471508ctil
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Ethanol; Wound Closure Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Pterygium surgery using alcohol 20% + wound closure by bare sclera technique
  Interventions: Procedure: pterygium surgery using alcohol 20% for tissue separation and bare sclera as wound closure technique
- 2 (Active Comparator): Alcohol 20% for pterygium separation + wound closure by sliding flap technique.
  The main steps of surgery are described below.Wound closure technique is as follows.
  Disection of conjunctiva adjascent to the wound, bringing the dissected conjunctiva to the wound area and suturing by vicril 6/0 sutures
  Interventions: Procedure: pterygium surgery using alcohol 20% for tissue separation and bare sclera as wound closure technique
- 3 (Active Comparator): Alcohol 20 % for pterygium separation + using amniotic membrane and biological glue for wound closure.
  The steps of surgery are as described below, wound closure technique is as follows.
  Amniotic membrane is applied with its mesenchimal side to conjunctiva and glued by biological glue (main ingradients: calcium and thrombin)
  Interventions: Procedure: pterygium surgery using alcohol 20% for tissue separation and bare sclera as wound closure technique

INTERVENTIONS:
Procedure: pterygium surgery using alcohol 20% for tissue separation and bare sclera as wound closure technique — The eye operated is disinfected and covered according routine protocol.
  Tightly applying well above the pterygium area. Instilling alcohol 20% into the well and holding for 40-60 seconds. Absorbing alcohol by applicator and abundant irrigation with BSS.
  Pterygium separation starting 2 mm centrally from the edges of the tissue. Excising the pterygium tissue at the base. Applying mytomycin C for 2.5 min+ abundant irrigation with BSS.
  Wound closure by by technique described in each arm.
  Bandage with chloramphenicol ointment or with Maxitrol ointment (Dexamethasone/Neomycin/Polymyxin B Eye Ointment.
  Postoperative treatment include :antibiotic and steroid eyedrop treatment at least 2 weeks.
  Follow up at 1 week, 1 month, 3 months, 6 months, 1 year. If additional follow upvisits are needed - they will be accomplished according the patients condition and needs.

SUMMARY:
Purpose of this study is to evaluate efficiency and safety of Alcohol 20% for peeling pterygium and to compare 3 different methods of operative wound closure: Bare sclera, Sliding flap, Amniotic membrane + biological glue

DETAILED DESCRIPTION:
Pterygium is a fibrovascular tissue growing on conjunctiva and cornea. The disturbance/morbidity caused by pterygium is diverse, ranging from mild esthetic disturbance and till recurrent inflammations and significant decrease of visual acuity. Rate of pterygium is between 20%-49% of general population, while increase in these numbers is observed in the population of equatorial regions. Pterygium usually appears at age of 22-49 years. While the rate of pterygium appearance increases with the age, the recurrence rate after surgical removal is higher in younger patients. Treatment of pterygium is surgical. The main challenges during surgery are peeling of pterygium and prevention of recurrence. During the last two decades several methods were developed and became widely accepted for pterygium surgery. The emphasis in modifying pterygium surgery is done on initial phase of surgery - techniques of pterygium separation and the final phase - the wound closure methods, additionally adjuncts (such as Mitomycine C) became widely used. These modifications are considered to improve the surgical outcomes and decrease the rate of complications and recurrence rate. Currently popular techniques of pterygium separation include Blunt dissection + keratectomy (blunt separation of the tissue + dissection of superficial layers of cornea); Avulsion technique (Avulsion of the pterygium head by creating tension on the cap edge+ further optional blunt dissection); Air assisted dissection (injection of air into the side of pterygium cap to create good separation plane).

Alcohol 20% is widely used in surface refractive surgery, where it helps to peel easily the epithelium of the cornea. Several reports show a positive role of alcohol in treatment of recurrent corneal erosions resistant to other treatments. At microscopic level - the ethanol splits basement membrane at the level between lamina lucida and lamina densa, additionally ethanol destroys the hemidesmosome junctions between epithelial cells. No consensus exists on ethanol influence on keratocyte viability and function: some studies show delayed wound healing and significant keratocyte damage, while other works show no significant alteration in keratocyte number while using alcohol.

At the phase of pterygium separation our purpose is to check the safety and efficiency of alcohol 20% for peeling of pterygium from ocular surface.

Various closure techniques exist, 3 of the widespread techniques are: Bare sclera (with adjunct such as mitomycine C) - the wound is left as it is, without closure. Sliding conjunctival flap- conjunctiva from adjacent region is dissected, moved to the wound area and sutured. Amniotic membrane transplantation, using biological glue to adhere the membrane. Amniotic membrane does not carry HLA antigens - so that no HLA compatibility tests are needed. Amniotic membrane underwent screening of infectious diseases and was cryopreserved. Amniotic membrane is applied with its mesenchimal part towards sclera and basement membrane side upwards. Adhesion of amniotic membrane is achieved by biological glue (containing thrombin and calcium as main ingredients)

We intend to compare each of these methods of wound closure in conjunction with using alcohol 20 % for pterygium separation.

ELIGIBILITY:
Inclusion Criteria:

* Age- above 18 years old.
* Primary pterygium.
* Eligibility to sign the informed consent.

Exclusion Criteria:

* Unwillingness to participate in study.
* Hypersensitivity to materials/ medications used during the surgery.
* Pregnancy.
* Cases when the eye which should be operated is the only fuctional eye.
* Age less than 18 years old.
* Recurrent pterygium.
* Chronic eye diseases, especially ocular surface disorders such as: OCP, severe blepharitis, severe keratoconjunctivitis,atopic eye disorders.

Patients which are not eligible to sign independently the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | during first 3 months
pterygium recurrence | at least 1 year

SECONDARY OUTCOMES:
patient satisfaction | during 1 year
corneal topography | during 1 year
endothelial cell density | during 1 year
evaluation of risk factors for pterygium recurrence (ex. exposure to UV-light, family history ...) | during 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tova Lifshitz, MD, Principal Investigator — Professor, Chief of ophthalmology department and clinics, SorokaUniversity Medical Center, Israel
Locations (2):
- Israel (2):
  - Soroka University Medical Center, Ophthalmology department and outpatient clinics, Beersheba
  - Soroka University Medical Center, Beersheba